CLINICAL TRIAL: NCT01798992
Title: Beta-blocker Effect on Structural Remodeling and Gene Expression in the Failing Human Heart
Brief Title: Effect of Beta-blockers on Structural Remodeling and Gene Expression in the Failing Human Heart
Acronym: BORG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); GlaxoSmithKline (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 00-0242; 2R01HL048013 (NIH)
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Idiopathic Dilated Cardiomyopathy
Keywords: ejection fraction; beta-blocker; carvedilol; metoprolol; myocardial gene expression; human heart; ventricular remodeling; wall stress; adrenergic signaling; myosin heavy chain
MeSH Terms: conditions — Cardiomyopathy, Dilated; Ventricular Remodeling | interventions — Carvedilol; Metoprolol; Doxazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Non-failing control (No Intervention): Patients with normal ejection fraction who underwent a single myocardial biopsy and received no β-blocker therapy
- Metoprolol succinate (Active Comparator): Idiopathic dilated cardiomyopathy patients randomized to metoprolol succinate titrated to a goal of 200 mg by mouth daily for 18 months
  Interventions: Drug: Metoprolol succinate
- Metoprolol succinate + doxazosin (Active Comparator): Idiopathic dilated cardiomyopathy patients who were randomized to receive metoprolol succinate and doxazosin titrated to a goal of 200 mg and 8 mg by mouth daily for 18 months
  Interventions: Drug: Metoprolol succinate + doxazosin
- Carvedilol (Active Comparator): Idiopathic dilated cardiomyopathy patients who were randomized to receive carvedilol titrated to a goal of 25 mg by mouth twice daily for 18 months
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol
  Other Names: Coreg
  Arms: Carvedilol
Drug: Metoprolol succinate
  Other Names: Toprol XL
  Arms: Metoprolol succinate
Drug: Metoprolol succinate + doxazosin
  Other Names: Toprol XL; Cardura; Carduran
  Arms: Metoprolol succinate + doxazosin

SUMMARY:
The primary goal of the study is to measure in the intact human heart, the alterations in gene expression over time that are associated with reverse remodeling in response to β-blockade. The second goal is to investigate the signaling mechanisms which in turn are responsible for these changes in gene expression, and the third goal is to determine the relationship between intrinsic systolic dysfunction and remodeling of the left ventricle. This will be accomplished by measuring ventricular size, function, and gene expression in myocardial tissue samples obtained by percutaneous biopsy prior to initiation of β-blockade and at 3 and 12 months after start of therapy. The specific Aims and Hypotheses to be tested are:

1. Aim: Determine the changes in gene expression associated with changes in intrinsic systolic function and with functional decompensation in the intact, failing human heart.

   a. Hypothesis: Changes in the expression of select genes precede or accompany changes in left ventricular systolic function in humans with idiopathic dilated cardiomyopathy (IDC).
2. Aim: Identify signaling mechanisms responsible for alterations in expression of key genes involved in mediation of ventricular hypertrophy or contractile dysfunction.

   a. Hypothesis: Myocardial-failure-associated regulation of select messenger ribonucleic acids and proteins are related to left ventricular wall stress and neurohormonal signaling.
3. Aim: In the relationship between contractile dysfunction and dilatation/remodeling, determine the relationship between contractile dysfunction and structural remodeling.

   b. Hypothesis: the contractile dysfunction is primary and structural remodeling secondary.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic dilated cardiomyopathy with New York Heart Association Class II-IV symptoms
* No evidence of coronary artery disease by angiography within 2 years of randomization
* If female, patient is (a) surgically sterile or (b) practices an accepted method of birth control and has negative serum pregnancy test
* Patient has been on other conventional cardiac heart failure(CHF) therapy at least 3 weeks prior to baseline assessments (includes angiotensin converting enzyme inhibitors, digoxin, diuretics, and/or vasodilators)
* Patient has left ventricular ejection fraction < 40% by radionuclide ventriculography within 60 days of randomization
* Patient must demonstrate mental and physical ability and willingness to follow all study-specific instructions
* Patient must voluntarily sign Institutional Review Board (IRB)-approved informed consent form prior to any study-specific procedure

Exclusion Criteria:

* Patient has heart failure due to or associated with uncorrected primary valvular disease, uncorrected thyroid disease, obstructive/hypertrophic cardiomyopathy, pericardial disease, amyloidosis, active myocarditis, or malfunctioning artificial heart valve.
* Patient is actively on heart transplant list or anticipated to be within 6 months of randomization
* Patient is receiving any of the following medicines:

  1. Calcium channel blockers
  2. Theophylline
  3. Tricyclic antidepressants
  4. Monoamine oxidase inhibitors
  5. β-agonists
  6. β-adrenergic blocking agent (oral)
  7. Any investigational cardiovascular medication or involvement in another investigational trial
  8. Flecainide, encainide, propafenone, sotalol, disopyramide, or amiodarone
* Patient has a contraindication to β-blockade (eg asthma)
* Patient has another life-threatening disease with life expectancy < 2 years due to other illness
* Patient has active hepatic, renal, hematologic, gastrointestinal, immunologic, endocrine, metabolic, or central nervous system disease which may adversely affect the safety and efficacy of the study drug or life span of the patient
* Unstable decompensated heart failure (evidence of hypoperfusion, acute pulmonary edema, or hypotension with SBP < 80 mm Hg)
* Patient is actively abusing ethanol or illicit drugs within 3 months of randomization
* Patient has an automatic implantable cardiac defibrillator that has fired within 3 months of randomization
* Patient has an asymptomatic waking, resting heart rate < 50 bpm or symptomatic bradycardia < 60 bpm.
* Patient has uncontrolled insulin-dependent diabetes mellitus with a history of frequent hypoglycemia episodes
* Patient has a high degree atrioventricular block (Mobitz Type II or complete heart block)
* Patient is unable to tolerate magnetic resonance imaging procedures
* Patient has demonstrated non-compliance with previous medical regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2000-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Bristow, MD PhD, Principal Investigator — University of Colorado School of Medicine
Locations (2):
- United States (2):
  - University of Colorado Hospital, Denver, Colorado
  - University of Utah Medical Center, Salt Lake City, Utah

REFERENCES:
- [Derived] Sucharov CC, Kao DP, Port JD, Karimpour-Fard A, Quaife RA, Minobe W, Nunley K, Lowes BD, Gilbert EM, Bristow MR. Myocardial microRNAs associated with reverse remodeling in human heart failure. JCI Insight. 2017 Jan 26;2(2):e89169. doi: 10.1172/jci.insight.89169. PMID 28138556
- [Derived] Kao DP, Lowes BD, Gilbert EM, Minobe W, Epperson LE, Meyer LK, Ferguson DA, Volkman AK, Zolty R, Borg CD, Quaife RA, Bristow MR. Therapeutic Molecular Phenotype of beta-Blocker-Associated Reverse-Remodeling in Nonischemic Dilated Cardiomyopathy. Circ Cardiovasc Genet. 2015 Apr;8(2):270-83. doi: 10.1161/CIRCGENETICS.114.000767. Epub 2015 Jan 30. PMID 25637602

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between 9/1/2000 and 3/1/2008 from outpatient general cardiology and heart failure specialty clinics at the University of Colorado Hospital and University of Utah Health Sciences Center.
Pre-assignment Details: 65 patients met screening criteria and provided consent. Exclusions included personal preference (4), administrative reasons such as relocation (2), normalization of LVEF prior to assignment (2), and lack of central venous access (1).
Groups:
- Metoprolol Succinate: Idiopathic dilated cardiomyopathy patients randomized to metoprolol succinate titrated to a goal of 200 mg by mouth daily for 18 months
  Metoprolol succinate
- Metoprolol Succinate + Doxazosin: Idiopathic dilated cardiomyopathy patients who were randomized to receive metoprolol succinate and doxazosin mesylate titrated to goals of 200 mg (metoprolol succinate) and 8 mg (doxazosin mesylate) by mouth daily for 18 months
  Metoprolol succinate + doxazosin
- Carvedilol: Idiopathic dilated cardiomyopathy patients who were randomized to receive carvedilol titrated to a goal of 25 mg by mouth twice daily for 18 months
  Carvedilol
Period: Overall Study
Arm/Group | Non-failing Control | Metoprolol Succinate | Metoprolol Succinate + Doxazosin | Carvedilol
Started | 4 | 19 | 16 | 17
Completed | 4 | 17 | 14 | 16
Not Completed | 0 | 2 | 2 | 1
Not completed — Administrative withdrawal | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Insufficient biopsy tissue | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients who gave informed consent and underwent baseline imaging and endomyocardial biopsy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-failing Control | Metoprolol Succinate | Metoprolol Succinate + Doxazosin | Carvedilol | Total
Number analyzed (Participants) | 4 | 19 | 16 | 17 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] — Calculated using enrollment date - birthdate
  years | 41.0 (17.1) | 45.9 (13.6) | 46.0 (7.5) | 44.9 (15.1) | 45.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 6 | 5 | 16
  Male | 3 | 15 | 10 | 12 | 40
Race/Ethnicity, Customized [Number; unit: participants]
  European Ancestry | 4 | 15 | 9 | 13 | 41
  African Ancestry | 0 | 1 | 4 | 0 | 5
  Hispanic | 0 | 2 | 1 | 4 | 7
  Other | 0 | 1 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 19 | 16 | 17 | 56
LV ejection fraction [Mean (Standard Deviation); unit: %] — Left ventricular ejection fraction = Stroke volume/End diastolic volume. Measured by single-photon emitted computed tomographic (SPECT) imaging or where not available, clinical multi-gated acquisition (MUGA) radionuclide ventriculography
  % | 58.8 (7.4) | 22.5 (7.1) | 28.5 (8.7) | 28.6 (8.7) | 28.6 (11.9)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Left Ventricular Ejection Fraction (LVEF) at 12 Months
Description: The primary clinical outcome will be LVEF response at 12 months defined as an improvement in LVEF of ≥ 8% at 12 months or if not available, ≥5% at 3 months in the absence of an adverse clinical outcome. Data are not presented for non-failing controls, who only went baseline evaluation and did not undergo treatment, given that they did not have heart failure.
Time Frame: 12 months
Population: Idiopathic dilated cardiomyopathy patients naive to beta-blocker therapy
Measure: Number; unit: LVEF responders
Groups:
- Metoprolol Succinate + Doxazosin: Idiopathic dilated cardiomyopathy patients who were randomized to receive metoprolol succinate and doxazosin titrated to a goal of 200 mg and 8 mg by mouth daily for 18 months
  Metoprolol succinate + doxazosin
Arm/Group | Metoprolol Succinate | Metoprolol Succinate + Doxazosin | Carvedilol
Number analyzed (Participants) | 17 | 14 | 16
LVEF responders | 12 | 10 | 9
Statistical Analysis 1: Comparison: Metoprolol Succinate vs Metoprolol Succinate + Doxazosin vs Carvedilol; The null hypothesis is that there is no difference in rate of LVEF improvement according to treatment group; Test type: Superiority or Other; p = 0.685, Fisher Exact

2. Secondary Outcome: Improvement in LVEF at 3 Months
Description: A secondary outcome will be LVEF response at 3 months, defined as an improvement of ≥ 5% Data are not presented for non-failing controls, who only went baseline evaluation and did not undergo treatment, given that they did not have heart failure.
Time Frame: 3 months
Measure: Number; unit: LVEF responders
Arm/Group | Metoprolol Succinate | Metoprolol Succinate + Doxazosin | Carvedilol
Number analyzed (Participants) | 17 | 14 | 16
LVEF responders | 16 | 10 | 10
Statistical Analysis 1: Comparison: Metoprolol Succinate vs Metoprolol Succinate + Doxazosin vs Carvedilol; The null hypothesis is that there is no difference in rate of LVEF improvement according to treatment group; Test type: Superiority or Other; p = 0.071, Fisher Exact

3. Secondary Outcome: Composite of All-cause Mortality, Need for Heart Transplant or Need for Ventricular Assist Device.
Description: Clinical status at 18 months will be assessed at time of study completion, specifically for the composite outcome of all-cause mortality, need for heart transplant, or need for ventricular assist device. Outcomes are not presented for non-failing controls, who only went baseline evaluation and did not undergo treatment, given that they did not have heart failure.
Time Frame: 18 months
Population: Idiopathic dilated cardiomyopathy patients randomized to different beta-blocker strategies. Data does not include non-failing controls, as these patients only underwent baseline evaluation with no treatment or follow-up, given that they did not have heart failure.
Measure: Number; unit: participants
Arm/Group | Metoprolol Succinate | Metoprolol Succinate + Doxazosin | Carvedilol
Number analyzed (Participants) | 17 | 14 | 16
participants | 1 | 0 | 0

4. Other Pre Specified Outcome: Change in Myocardial Gene Expression at 3 Months
Description: Changes in myocardial mRNA expression at 3 months compared to baseline using targeted quantitative polymerase chain reaction and genome wide microarray assays. Due to the large number of results genes interrogated (~ 20,000 genes), these results will instead be uploaded to the Gene Expression Omnibus.
Time Frame: 3 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Myocardial Gene Expression at 12 Months
Description: Changes in myocardial mRNA expression at 12 months compared to baseline using targeted quantitative polymerase chain reaction and Affymetrix genome-wide microarray assays. Data are not presented for non-failing controls, who only went baseline evaluation and did not undergo treatment, given that they did not have heart failure.
Time Frame: 12 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Myocardial microRNA Expression at 3 Months
Description: Changes in myocardial microRNA expression at 3 months compared to baseline using an Affymetrix microRNA microarray assay. Data are not presented for non-failing controls, who only went baseline evaluation and did not undergo treatment, given that they did not have heart failure.
Time Frame: 3 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Myocardial microRNA Expression at 12 Months
Description: Changes in myocardial microRNA expression at 12 months compared to baseline using an Affymetrix microRNA microarray assay. Data are not presented for non-failing controls, who only went baseline evaluation and did not undergo treatment, given that they did not have heart failure.
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Metoprolol Succinate | Metoprolol Succinate + Doxazosin | Carvedilol
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/14 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No